CLINICAL TRIAL: NCT06222671
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase II Clinical Study to Evaluate the Efficacy and Safety of 608 in Patients With Non-radiographic Axial Spondyloarthritis (Nr-axSpA)
Brief Title: A Study to Evaluate 608 in Patients With Non- Radiographic Axial Spondyloarthritis (Nr-axSpA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-608-nr-axSpA-II-01
Record Dates: First submitted 2024-01-10; First posted 2024-01-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Axial Spondyloarthritis
Keywords: non-radiographic axial spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis; Non-Radiographic Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 608 Dose A (Experimental): 608 Dose A subcutaneous (SC) injection.
  Interventions: Drug: 608
- 608 Dose B (Experimental): 608 Dose B subcutaneous (SC) injection.
  Interventions: Drug: 608
- Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 608 — 608 subcutaneous (SC) injection.
  Arms: 608 Dose A
Drug: 608 — 608 subcutaneous (SC) injection.
  Arms: 608 Dose B
Drug: Placebo — Placebo subcutaneous (SC) injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the effect and safety of 608 in patients with nr-axSpA.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the clinical efficacy, safety and tolerability of 608 compared to placebo in patients with nr-axSpA.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients at least 18 years of age at the time of screening.
2. Diagnosis of axial spondyloarthritis according to Ankylosing Spondylo Arthritis International Society (ASAS) axial spondyloarthritis criteria
3. Objective signs of inflammation (magnetic resonance imaging (MRI) or abnormal C-reactive protein)
4. Total back pain as measured by NRS ≥ 4 at baseline

Exclusion Criteria:

1. Patients with other uncontrolled active inflammatory diseases.
2. Clinical laboratory tests and other tests that reveal abnormalities with clinical significance
3. Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
4. History of cancer.
5. Known or suspected history of immunosuppression.
6. Known with allergic or intolerant to mometasone furoate spray or 608/placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 40 Response | From Baseline to Week 16
  Assessment of Spondylo Arthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the NRS signifies higher severity.

SECONDARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 20 Response | From Baseline to the Week 16
  Assessment of Spondylo Arthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS 20 response is defined as an improvement of ≥20% and ≥1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain. A higher score on the NRS signifies higher severity.
608 Concentration in Serum | From Baseline to Week 24
  The concentration of 608 in Serum.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghong Zhou, BS, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.; Xiaofeng Zeng, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (6):
- China (6):
  - Site 01, Beijing, Beijing Municipality
  - Site 03, Beijing, Beijing Municipality
  - Site 05, Chongqing, Chongqing Municipality
  - Site 02, Zhengzhou, Henan
  - Site 04, Nanjing, Jiangsu
  - Site 06, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No